CLINICAL TRIAL: NCT07327021
Title: NOGA: Neoadjuvant Treatment Optimization Via MRI-Guided De-Escalation in Stage II-III TNBC - A Phase 2 Study.
Brief Title: MRI-Guided Neoadjuvant Treatment De-Escalation in Stage II-III TNBC
Acronym: NOGA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0369-25; 2347-25-SMC (Other: Sheba Medical Center)
Record Dates: First submitted 2025-11-20; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: TNBC, Triple Negative Breast Cancer; Early Breast Cancer
Keywords: TNBC; KEYNOTE-522; MRI
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Recruited patients will receive the first phase of the KEYNOTE-522 protocol (TCa+P). Breast MRI will be performed at baseline and repeated upon completion of the TCa+P phase. Patients demonstrating a complete response on MRI (MRI-CR) following 4 cycles of TCa+P will be referred for early surgery. Patients with residual disease on MRI (MRI-RD) will complete the KEYNOTE-522 regimen with up to four 21-day cycles of AC+P.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI Complete Response (MRI-CR) (Experimental): Radiological complete response in MRI after the first phase of the KEYNOTE-522 regimen (TCa+P)
  Interventions: Other: Treatment De-Escalation and Early Surgery
- MRI Residual Disease (MRI-RD) (No Intervention): Radiological residual disease in MRI after the first phase of the KEYNOTE-522 regimen (TCa+P)

INTERVENTIONS:
Other: Treatment De-Escalation and Early Surgery — Patients with MRI-CR after the first phase of the KEYNOTE-522 regimen will be referred for early surgery without completing the AC+P phase.
  Arms: MRI Complete Response (MRI-CR)

SUMMARY:
Breast cancer is the most common malignancy among women worldwide. Triple-negative breast cancer (TNBC), defined by the lack of estrogen receptor, progesterone receptor, and HER2 expression, comprises approximately 15% of all breast cancers and is the most aggressive subtype, associated with a higher risk of early recurrence and death compared to other breast cancer subtypes. Neoadjuvant chemotherapy (NACT), administered before definitive surgery, is the standard of care for stage II-III TNBC (eTNBC), and pathological complete response (pCR), defined as the absence of invasive cancer in the breast and lymph nodes at surgery, following neoadjuvant systemic therapy, is strongly associated with improved survival in this population.

In the pivotal phase 3 KEYNOTE-522 study, the addition of Pembrolizumab (an immune checkpoint inhibitor (ICI), a PD-1 inhibitor) to NACT significantly improved both pCR rates and survival in patients with eTNBC , establishing a new standard of care for these patients. The KEYNOTE-522 regimen is a five-drug regimen administered in two distinct phases: in the first phase, Paclitaxel and Carboplatin are administered with Pembrolizumab for four cycles (TCa+P) and in the second phase, Adriamycin and Cyclophosphamide are administered with Pembrolizumab for an additional four cycles (AC+P). This regimen carries a high toxicity burden, particularly due to anthracyclines, which are associated with late cardiotoxicity and increased risk of therapy-related leukemias.

Many patients, however, achieve an excellent response after only the first phase of treatment (paclitaxel-carboplatin + pembrolizumab), raising the question of whether treatment can be safely de-escalated in selected responders. Emerging evidence from the NeoPACT and NEO-N studies suggests that pCR rates of 55-58% can be achieved with taxane-carboplatin-pembrolizumab regimen, even in the absence of anthracyclines. Moreover, the recently published TRAIN-3 study in HER2+ breast cancer demonstrated that radiologic complete response on MRI (MRI-CR) strongly correlates with pCR in hormone receptor-negative disease, with 87% concordance.

Building on this rationale, we propose a prospective, investigator-initiated, multicenter, phase II clinical trial in Israel to evaluate the feasibility and efficacy of MRI-guided de-escalation of NACT plus immunotherapy in patients with eTNBC. All enrolled patients will receive four cycles (12 weeks) of paclitaxel-carboplatin with pembrolizumab (TCa+P), followed by breast MRI to assess treatment response. Patients achieving MRI-CR will proceed directly to surgery, omitting the second phase of anthracycline-containing chemotherapy (AC+P). Patients with radiologic residual disease (MRI-RD) will complete the full KEYNOTE-522 regimen. Adjuvant therapy, including pembrolizumab continuation and/or additional chemotherapy, will be administered based on pathological findings and physician and patient discretion.

The primary endpoint is pCR rate among patients who achieve MRI-CR and undergo early surgery. The trial uses a Simon's two-stage optimal design and aims to test whether the observed pCR rate in MRI-CR patients exceeds the benchmark of 65% (based on KEYNOTE-522), with a target of 87% as suggested by TRAIN-3. Based on this approach, to reject the null hypothesis, a pathologic complete response (pCR) must be achieved in at least 22 of the 27 patients with MRI-CR who are referred to early surgery. Overall, Approximately 54 patients will be enrolled in the study to reach this goal. Key secondary endpoints include recurrence-free survival (RFS), overall survival (OS), and patient-reported quality of life (QoL). Patient-reported outcomes (PROs) will be collected longitudinally throughout the study to assess physical symptoms, psychological well-being, treatment-related toxicities, and functional recovery, helping to evaluate how treatment de-escalation impacts patient's experience.

In addition, the study will prospectively collect blood samples for circulating tumor DNA (ctDNA) analysis, creating a unique biorepository of biologic material for translational research. ctDNA dynamics will be evaluated as a complementary biomarker to MRI, enabling assessment of early treatment response, molecular residual disease, and mechanisms of resistance. Samples will be collected at multiple timepoints, before treatment, during therapy, and prior to surgery, providing a rich dataset for future genomic, epigenetic, and immune profiling studies.

This study represents an innovative, precision-driven approach to treatment de-escalation in eTNBC, with the potential to influence clinical practice and redefine the standard of care by identifying patients who can safely avoid anthracycline-based chemotherapy without compromising efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible per physician's discretion for the KEYNOTE-522 regimen (Neoadjuvant paclitaxel-carboplatin-doxorubicin-cyclophosphamide-pembrolizumab)
* Signed written informed consent
* Histologically confirmed primary infiltrating breast cancer with estrogen receptor expression <1%, Progesterone receptor expression <1%, and without overexpression and/or amplification of HER2 according to ASCO/CAP 2013 guideline (locally assessed)
* T2-3N0, T1-3N1 disease according to TNM-staging (8th edition, AJCC).
* Nodal status must be examined by ultrasound and fine-needle aspiration or core biopsy in case of suspicious lymph nodes.
* No evidence of distant metastases (Stage IV disease) on FDG-PET performed within 35 days of enrollment.
* Age ≥18
* WHO performance status ≤ 2
* Visible breast tumor on contrast enhanced MRI (no minimal longest diameter required)
* MRI breast must be performed within 35 days prior to registration
* Patients with a history of autoimmune disease are eligible for the study per treating physician's discretion.
* Laboratory requirements - within 21 days prior to enrollment:

  * Adequate bone marrow function (ANC ≥1.5 x 109/l, platelets ≥100 x 109/l)
  * Adequate hepatic function (ALT, AST and bilirubin ≤2.5 times upper limit of normal)
  * Subjects with Gilbert's syndrome may have a total bilirubin ≥2.5 × the ULN range, if no evidence of biliary obstruction exists;
  * Adequate renal function: creatinine clearance >50 ml/min estimated using the Cockcroft-Gault equation, or based on a 24-hour urine collection measurement
  * LVEF ≥50% measured by echocardiography
* Women of childbearing potential and men must agree to remain abstinent (refrain from heterosexual intercourse) or use adequate contraceptive methods (failure rate of <1% per year,) during treatment and for at least 6 months after the last dose of pembrolizumab. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs. Women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative β-HCG serum or urine pregnancy test result.

Exclusion Criteria:

* Concurrent breastfeeding
* Concurrent contralateral or ipsilateral non-TNBC second primary infiltrating breast cancer. Contralateral or ipsilateral TNBC second primary infiltrating breast cancer or DCIS is allowed.
* Concurrent anti-cancer treatment or another investigational drug
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Patients who have a history of a second malignancy are eligible, provided the malignancy has been adequately treated, there is no ongoing treatment for the second malignancy, and overall principal investigator (PI) approval is obtained.
* Has undergone excisional biopsy of the primary tumor, and/or axillary lymph node dissection prior to study treatment.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's ability to cooperate with the requirements of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate in patients with MRI-CR following TCa+P treatment who proceeded to early surgery | up to 24 weeks
  pCR in breast and axilla, defined as the absence of invasive tumor cells, irrespective of the presence of in-situ lesions.

SECONDARY OUTCOMES:
Recurrence Free Survival (RFS) rate, as assessed by Kaplan-Meier method | up to 3 years
  Percentage of patients with RFS as assessed by Kaplan-Meier method. Recurrence-free survival (RFS) in the MRI-CR group and in all patients. RFS defined as the interval from registration to the earliest occurrence of disease progression resulting in inoperability, invasive loco regional recurrence, distant metastases, or death from any cause, whichever comes first.
Overall Survival (OS) rate, as assessed by Kaplan-Meier method | Up to 3 years
  OS as assessed by Kaplan-Meier method. OS is defined as the length of time from randomization until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No